CLINICAL TRIAL: NCT02688777
Title: A Novel Strategy to Decrease Fall Incidence Post-Stroke
Acronym: BLAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N2004-R
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Rehabilitation; Gait; Postural Balance; Exercise; Accidental Falls; Kinesiology, Applied
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel: participants are assigned to one of two or more groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Backward Walking Training (Experimental): Individuals will participate in 18 sessions of Backward Walking training immediately following baseline assessment.
  Interventions: Behavioral: Backward Walking Training
- Delayed Backward Walking Training (Active Comparator): Individuals will participate in 18 sessions of Backward Walking training at 1-year post-strokeD
  Interventions: Behavioral: Backward Walking Training

INTERVENTIONS:
Behavioral: Backward Walking Training — Backward Walking Training will occur both on a treadmill and overground. In brief, BWTraining will consist of 20-30 minutes of step training with a Body Weight Support and Treadmill system (BWST), rest periods provided as warranted, with manual assistance provided by trainers, followed by 15 minutes of overground gait training. A 20-30 min period of actual stepping is the goal for the intervention sessions on the treadmill with rest periods as needed. Each training session may last up to 1 hour and 30 minutes including time for warm-up, stretching, and cool down. Participants will be fitted with a harness around their hips and torso, which will be attached to an overhead support system directly above the treadmill. From a stationary position, the treadmill belt will gradually be increased in speed with intervention trainers assisting participant to step backward with their paretic leg, their non-paretic leg (if needed) and at the hips for weight-shift.

SUMMARY:
Approximately 15,000 Veterans are hospitalized for stroke each year with new cases costing an estimated $111 million for acute inpatient, $75 million for post-acute inpatient, and $88 million for follow-up care over 6 months post-stroke. Contributing to these costs is the incidence of falls. Falls are a costly complication for Veterans with stroke as they lead to an increased incidence of fractures, depression, and mortality. New strategies are needed to help Veterans post-stroke regain their ability to safely walk without increasing their risk of falling as well as readily identify those who are a fall risk. This study addresses both of these needs as it will 1) investigate a new treatment approach, backward walking training, to determine if it will decrease fall incidence in the first year post-stroke and 2) determine if backward walking speed early after a stroke can identify those that are at risk for future falls.

DETAILED DESCRIPTION:
Approximately 15,000 Veterans are hospitalized for stroke each year. Persistent walking and balance deficits contribute to long-term disability and a high incidence of falls. Falls are a common and costly complication of stroke; between 40% and 70% of affected individuals fall within the first year. Falls lead to fear of falling, limitations in self-care and increased dependence. Of greater concern, they lead to serious adverse events, including fractures, depression and mortality. A primary goal of stroke rehabilitation is to improve mobility despite persistent motor, balance and visual-spatial deficits. However, this goal has a down side since it increases fall risks. Here, the investigators propose a novel therapeutic strategy to improve ambulation while decreasing the risk of falls: Backward Walking Training (BWTraining).

The investigators' central hypothesis is that a 6-week BWTraining program at 2-months post-stroke is superior to standard care in reducing falls within the 1st year post-stroke. Identification of those at risk for falling is a necessary component of post-stroke rehabilitation to implement pro-active measures to decrease risk once individuals rejoin community living. Recent research in a cohort of elderly adults determined that maximal Backward Walking Speed (BWSpeed) (not forward) identified individuals that had experienced a fall in the previous six months,6 suggesting that BWSpeed could be a simple, inexpensive screening tool to identify individuals at risk of falling. With a randomized, blinded design, the investigators propose to prospectively assess the value of BWSpeed as a tool to predict future falls.

A notable post-stroke conundrum is that increased mobility may increase fall risk.5 On the other hand, limiting mobility leads to a multitude of inactivity-associated deficits, including recurrent stroke.

To date, no intervention has demonstrated efficacy for improving walking while minimizing fall risk. BWTraining may be a simple and effective intervention to achieve both goals. In the investigators' recent randomized controlled pilot trial (RCT), individuals with sub-acute stroke who participated in a BWTraining demonstrated 3-fold improvement in backward and forward walking speed and fall self-efficacy. Further, BWTraining caused 75% greater improvement in balance versus those in a dose-matched balance training group. At the 3-month follow-up assessment, BWSpeed of the BWTraining group averaged 0.63 m/s, exceeding the threshold for fall risk in elderly adults.

Given the success of the investigators' pilot intervention, a larger and more rigorous trial is needed to demonstrate reduced fall incidence over an extended follow-up period. The investigators designed this RCT to address three specific aims:

Aim #1: Test the hypothesis that 1-year fall incidence is decreased for participants randomized to BWTraining administered at 2-months post-stroke (versus usual care comparison group).

Hypothesis #1a: BWTraining at 2-months post-stroke reduces the number of falls over the next year.

Hypothesis #1b: BWTraining at 2-months post-stroke increases gait speed, improves balance and increases balance confidence over the next year.

Aim #2: Test the hypothesis that BWTraining at 2 months (immediate) vs. 1-year (delayed) post-stroke is more effective at improving BWSpeed.

Hypothesis #2a: BWSpeed improvement from 2- to 14-months post-stroke is greater when BWTraining is delivered at 2 months versus 1 year post-stroke.

Hypothesis #2b: Improvements in forward gait speed, Functional Gait Assessment and Activities-Balance Confidence Scale from 2- to 14-months post-stroke are greater when BWTraining is delivered at 2 months versus 1 year post-stroke.

Aim #3: This exploratory aim will test the hypothesis that BWSpeed at 2-months post-stroke is a significant predictor of fall incidence over the next year 1 year period, after adjusting for other covariates.

Hypothesis #3: BWSpeed at 2-months will be a significant predictor of fall incidence during the first year post-stroke, after adjusting for other covariates.

This study is significant since it concerns a novel strategy to improve ambulation while minimizing the risk of falling after a stroke. BWTraining is highly novel, is easy to administer and exciting preliminary data suggest that is has major potential as a therapeutic tool. In addition, the investigators will determine the potential of BWSpeed (a simple, clinically relevant screening tool) to identify those at risk for future falls.

ELIGIBILITY:
Inclusion Criteria:

* Berg Balance Scale < 42
* Self-selected 10 meter gait speed < 0.8 m/s
* Diagnosis of unilateral stroke
* > 2 months < 4 months post-stroke
* Able to ambulate at least 10 feet with maximum 1 person assist
* Medically stable
* 18-85 years of age
* Physician approval for patient participation

Exclusion Criteria:

* Presence of neurological condition other than stroke
* Serious cardiac conditions

  * hospitalization for myocardial infarction or heart surgery within 3 months
  * history of congestive heart failure
  * documented serious and unstable cardiac arrhythmias
  * hypertrophic cardiomyopathy
  * severe aortic stenosis
  * angina or dyspnea at rest or during activities of daily living
* Anyone meeting New York Heart Association criteria for Class 3 or Class 4 heart disease will be excluded
* Severe arthritis or orthopedic problems that limit passive ranges of motion of lower extremity

  * knee flexion contracture of -10
  * knee flexion Range Of Motion < 90
  * hip flexion contracture > 25
  * ankle plantar flexion contracture > 15
* Severe hypertension with systolic greater than 200 mmHg and diastolic greater than 110 mmHg at rest, that cannot be medically controlled into the resting range of 180/100 mmHg
* Pain upon ambulation
* Receiving physical therapy services for mobility and/or gait
* Living in a skilled nursing facility
* Unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking less than 200 meters
* History of serious chronic obstructive pulmonary disease or oxygen independence
* Non-healing ulcers on the lower extremity
* Uncontrollable diabetes with recent weight loss, diabetic coma or frequent insulin reactions
* On renal dialysis or presence of end stage liver disease
* Pulmonary embolism within previous 6 months
* History of major head trauma
* History of sustained alcoholism or drug abuse in the last six months
* Intracranial hemorrhage related to aneurysmal rupture or an arteriovenous malformation
* Current enrollment in a clinical trial to enhance stroke motor recovery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Kay Rose, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Backward Walking Training: Individuals will participate in 18 sessions of Backward Walking training immediately following baseline assessment.
  Backward Walking Training (BWTraining): Backward Walking Training will occur both on a treadmill and overground. In brief, Backward Walking Training (BWTraining) will consist of 20-30 minutes of step training with a Body Weight Support and Treadmill system (BWST), rest periods provided as warranted, with manual assistance provided by trainers, followed by 15 minutes of overground gait training. A 20-30 min period of actual stepping is the goal for the intervention sessions on the treadmill with rest periods as needed. Each training session may last up to 1 hour and 30 minutes including time for warm-up, stretching, and cool down. Participants will be fitted with a harness around their hips and torso, which will be attached to an overhead support system directly above the treadmill. From a stationary position, the treadmill belt will gradually be increased in speed with intervention trainers assisting participant to step backward with their paretic leg, their non-paretic leg (if needed) and at the hips for weight-shift.
- Delayed Backward Walking Training: Individuals will participate in 18 sessions of Backward Walking training at 1-year post-stroke
  Backward Walking Training: Backward Walking Training will occur both on a treadmill and overground. In brief, BWTraining will consist of 20-30 minutes of step training with a Body Weight Support and Treadmill system (BWST), rest periods provided as warranted, with manual assistance provided by trainers, followed by 15 minutes of overground gait training. A 20-30 min period of actual stepping is the goal for the intervention sessions on the treadmill with rest periods as needed. Each training session may last up to 1 hour and 30 minutes including time for warm-up, stretching, and cool down. Participants will be fitted with a harness around their hips and torso, which will be attached to an overhead support system directly above the treadmill. From a stationary position, the treadmill belt will gradually be increased in speed with intervention trainers assisting participant to step backward with their paretic leg, their non-paretic leg (if needed) and at the hips for weight-shift.
Period: Overall Study
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Started | 32 | 30
Completed | 25 | 19
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 20 | 44
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.8) | 57.8 (14.5) | 58.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 11 | 23
  White | 16 | 18 | 34
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Fall Incidence (Number of Falls)
Description: Fall incidence will be monitored using the international standards for defining and reporting falls,60 including the following definition for a fall: "A person has a fall if they end up on the ground or floor when they did not expect to. Most often a fall starts while a person is on their feet, but a fall could also start from a chair or bed. If a person ends up on the ground, either on their knees, their belly, their side, their bottom, or their back, they have had a fall." This explanation will be provided to participants and caregivers and printed on monthly calendars issued at randomization. The number of falls will be recorded on a monthly basis and then added across months to determine the number of recorded falls between baseline and 1-year post-stroke.
Time Frame: Number of recorded falls between baseline and 1-year post-stroke
Measure: Number; unit: number of falls
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
number of falls | 88 | 56
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; Hazard Ratio, log = 0.6

2. Secondary Outcome: 10 Meter Walk Test
Description: Individuals will be given a 2 meter warm-up distance for walking, preceding the 10 meter distance and 2 meters beyond the 10 meters to continue walking. The time that it takes to traverse the 10 meters at the subject's usual pace will be recorded.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: meters/second
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
meters/second | 0.17 (0.03) | 0.22 (0.04)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.37, t-test, 2 sided — A priori threshold for significance is p < 0.05; Mean Difference (Final Values) = 0.05, Standard Error of Mean 0.03

3. Secondary Outcome: 3-Meter Backward Walk Test
Description: The test consists of a 1 meter warm-up distance, a timed 3 meter distance, followed by an additional 1 meter to continue walking An average of two trials will be recorded.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
meters/second | 0.13 (0.02) | 0.19 (0.03)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.13, t-test, 2 sided — A priori threshold set for p < 0.05; Mean Difference (Final Values) = 0.16, Standard Error of Mean 0.02

4. Secondary Outcome: Functional Gait Assessment
Description: A 10-item clinical gait and balance test during which participants perform the following activities: walk at normal speeds, at fast and slow speeds, with vertical and horizontal head turns, with eyes closed, over obstacles, in tandem, backward and while ascending and descending stairs.
  Minimum value: 0 Maximum value: 40 Higher score = better outcome
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
score on a scale | 4.8 (0.84) | 5.6 (1.1)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.40, t-test, 2 sided — A priori threshold p < 0.05 for statistical significance; Mean Difference (Final Values) = 0.8, Standard Error of Mean 1.0

5. Secondary Outcome: Activities-Specific Balance Confidence Scale
Description: This 16-item self-report measure is used to assess perceived efficacy (self-reported confidence) in maintaining balance while performing a number of activities common in community-dwelling older adults.
  Minimum value: 0% Maximum value: 100% Higher score = better outcome
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: percentage of confidence
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
percentage of confidence | 15.9 (3.4) | 21.6 (3.5)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.12, t-test, 2 sided; Mean Difference (Final Values) = 5.7, Standard Error of Mean 3.4

6. Secondary Outcome: Berg Balance Scale
Description: This tool consists of 14 items that assesses static and dynamic standing balance, ability to sit, stand up and transfer.
  Minimum Value: 0 Maximum Value 56 Higher score = better outcome
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
score on a scale | 10.1 (1.8) | 10.4 (0.4)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.43, t-test, 2 sided — A priori threshold set at p < 0.05 for statistical significance; Mean Difference (Final Values) = 0.03, Standard Error of Mean 1.1

7. Secondary Outcome: Lower-Extremity Fugl-Meyer Motor Score
Description: This tool consists of 17 items that assess motor control of the lower extremity as participants move their hip, knee and ankle in lying, sitting and standing.
  Minimum score=0 Maximum score = 34 Higher score = better outcome
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
score on a scale | 2.6 (0.7) | 4.8 (0.9)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.02, t-test, 2 sided — A prior threshold for significance set at p < 0.05; Mean Difference (Final Values) = 2.2, Standard Error of Mean 0.8

8. Secondary Outcome: Four-Step Square Test
Description: This clinical test of dynamic standing balance examines the ability to step over small objects, change direction and includes taking a backwards step.
Time Frame: Change between baseline and 1-year post-stroke
Population: Not all participants were able to complete the Four Square Step Test. If the blinded assessor determined the participant would be unsafe completing this assessment, it was not conducted.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 28 | 23
seconds | 20.54 (6.89) | 34.49 (10.96)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = 13.95, Standard Error of Mean 8.9

9. Secondary Outcome: Stride Time
Description: Stride time will be captured during forward and backward walking across a pressure-sensitive instrumented walkway.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
seconds | 0.30 (0.03) | 0.26 (0.05)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 0.04

10. Secondary Outcome: Stride Length
Description: Stride length will be captured during forward and backward walking across a GAITRite instrumented walkway.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
centimeters | 5.1 (0.08) | 6.1 (0.09)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.10, t-test, 2 sided

11. Secondary Outcome: Step Time
Description: Step time will be captured during forward and backward walking across a GAITRite instrumented walkway.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
seconds | .116 (0.02) | .195 (0.03)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.09, t-test, 2 sided

12. Secondary Outcome: Step Length
Description: Step length will be captured during forward and backward walking across a GAITRite instrumented walkway.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
centimeters | 3.4 (1.2) | 5.0 (1.9)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.11, t-test, 2 sided

13. Secondary Outcome: Step Width
Description: Step width will be captured during forward and backward walking across a GAITRite instrumented walkway.
Time Frame: Change between baseline and 1-year post-stroke
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
Number analyzed (Participants) | 32 | 30
centimeters | 1.2 (0.06) | 2.2 (0.07)
Statistical Analysis 1: Comparison: Immediate Backward Walking Training vs Delayed Backward Walking Training; Test type: Superiority; p = 0.28, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Three years - over the course of the study.
Description: Monthly falls calendars were collected from participants.
Arm/Group | Immediate Backward Walking Training | Delayed Backward Walking Training
All-Cause Mortality (participants affected / at risk) | 0/32 | 1/30
Serious Adverse Events (participants affected / at risk) | 8/32 | 10/30
Other Adverse Events (participants affected / at risk) | 21/32 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Backward Walking Training (N=32) | Delayed Backward Walking Training (N=30)
Inpatient Hospitalization (General disorders) | 8 (14) | 10 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Backward Walking Training (N=32) | Delayed Backward Walking Training (N=30)
Fall without injury (General disorders) | 21 (87) | 18 (56)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT02688777/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT02688777/ICF_001.pdf